CLINICAL TRIAL: NCT06044857
Title: Phase IB Study of Personalized Ultrahypofractionated Stereotactic Ablative Radiotherapy of High Risk PROstate Cancer Guided by PET PSMA (68Ga PMSA-11; Ilucix) Response (PULSAR ProPhet)
Brief Title: PSMA PET Response Guided SabR in High Risk Pca
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Once Upon a Time Foundation (Other); Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Principal Investigator, Neil Desai, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0566
Record Dates: First submitted 2023-07-27; First posted 2023-09-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAbR Every other day (Experimental): SAbR given 2-3/week, at least every other day in spacing with long-term ADT (neoadjuvant ADT x 3months required) with experimental Illucix (PSMA-11 68Ga) PET before and during SAbR (between fraction 3 and 4) to assess and adapt to dominant intra-prostatic lesion boost dose.
  Interventions: Drug: 68-Ga PSMA11
- PULSAR every week (Experimental): SAbR given 1/week, with long-term ADT (neoadjuvant ADT x 3months required) with experimental Illucix (PSMA-11 68Ga) PET before and during SAbR (between fraction 3 and 4) to assess and adapt to dominant intra-prostatic lesion boost dose.
  Interventions: Drug: 68-Ga PSMA11
- PULSAR every 2 weeks (Experimental): SAbR given every 2 weeks, with long-term ADT (neoadjuvant ADT x 3months required) with experimental Illucix (PSMA-11 68Ga) PET before and during SAbR (between fraction 3 and 4) to assess and adapt to dominant intra-prostatic lesion boost dose.
  Interventions: Drug: 68-Ga PSMA11
- PULSAR every 3 weeks (Experimental): SAbR given every 3 weeks, with long-term ADT (neoadjuvant ADT x 3months required) with experimental Illucix (PSMA-11 68Ga) PET before and during SAbR (between fraction 3 and 4) to assess and adapt to dominant intra-prostatic lesion boost dose.
  Interventions: Drug: 68-Ga PSMA11

INTERVENTIONS:
Drug: 68-Ga PSMA11 — Will be injected/assessed in line with its FDA label.
  Other Names: Illucix, Telix

SUMMARY:
Sequential cohort evaluation of ideal timing of imaging and treatment spacing to discern maximal PSMA (Prostate specific membrane antigen) PET (Positron Emission Tomography) response (PSMA-11 68Ga, Illucix) for adaptation of dominant intra-prostatic lesion tumor boost dose

ELIGIBILITY:
Inclusion Criteria:

-Pathologically confirmed adenocarcinoma of the prostate (within 180 days of registration) of high risk by national comprehensive cancer network (NCCN) criteria as determined by >=cT3a stage (AJCC 8th edition) OR PSA>20ng/mL OR ISUP Grade Group 4-5 (Gleason Grade 8-10).

Age ≥ 18 years.

* Planned for definitive intent stereotactic ablative radiotherapy (SabR) with integrated dose boost to intra-prostatic tumor and androgen deprivation therapy (ADT) with baseline AUA IPSS <=18 and prostate size <=100cc
* Staging 68Ga PMSA-11 PET -CT or -MRI performed within 90 days of registration and before initiation of anti-androgen or androgen deprivation therapy and demonstrating no evidence of distant metastases by (PMSA avid or non-avid nodes <=1.5cm short axis allowed). Conventional imaging (CT, bone scan, MRI) may also be used in addition to PMSA-PET, and definitive findings of distant extra-pelvic metastases on these scans are not allowed for enrollment.
* Staging 68Ga PSMA-11 PET -CT or -MRI demonstrating a PSMA-avid primary intra-prostatic target lesion amenable at investigator discretion to dose boost
* All men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of standard of care SabR and for a period of time of 6 months thereafter as per standard guidelines. Should a man's partner become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior curative intent local therapy (e.g. prostatectomy, radiotherapy, focal ablative therapy) for prostate cancer is not allowed, with following exceptions regarding androgen deprivation therapy (ADT)/anti-androgen therapy (AAT):

Prior androgen deprivation therapy (ADT) allowed if <3 month total duration and stopped >=3 months prior to registration with demonstration of non-castrate testosterone recovery (>50ng/dL) and meeting all other inclusion criteria.

Ongoing androgen deprivation therapy (ADT) is allowed if <=60 days total duration AND meeting following criteria:

If GnRH agonist used (e.g. leuprolide), bicalutamide must have been used for at least 30 days +/-14 days from start of GnRH agonist.

All other inclusion criteria.

* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* History of allergic reactions to PMSA-11 68Ga imaging agent.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* Prior pelvic radiotherapy other than cutaneous/superficial treatments.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Target Intra-Prostatic Lesion(s) | Through end of neoadjuvant ADT at 3 months
  This study primarily evaluates volume reduction of initial target PSMA-avid dominant intra-prostatic disease after neoadjuvant ADT and during SAbR in differing spacing regimens of SAbR.
  Metrics include percent reduction in volume at 3 months of therapy vs initial disease extent of intra-prostatic dominant lesion as identified by PSMA PET.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Desai, MD MHS, Principal Investigator — Study Principal Investigator
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided